CLINICAL TRIAL: NCT07362056
Title: Integrating a Suicide Prevention Package of Strategies Into Decentralized Primary Health Care Systems: an Implementation Pilot Study in Rural Nepal
Brief Title: Implementing Suicide Prevention Into Primary Care in Nepal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Possible (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000036105; 5R34MH135122 (NIH); 1R34MH135122-01 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Primary Care
Keywords: suicide prevention; primary care; implementation science; Nepal
MeSH Terms: conditions — Suicide; Suicide Prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): PCPs will receive standard or refresher mhGAP training. The training follows Nepal's district mental health plan for primary care workers with prescribing credentials. Paramedical staff are included because most primary healthcare facilities lack doctors, making them the primary frontline primary care providers. The training is based on the WHO mhGAP Intervention Guide and focuses on five priority conditions in Nepal: depression, psychosis, epilepsy, alcohol use disorder, and suicide. Training is delivered over 5 days by a Nepali psychiatrist with government issued credentials to facilitate mhGap training and subsequent ongoing supervision. After training, PCPs receive psychiatric supervision approximately every three months as per the Nepal government mhGap protocol. Patient participants in the TAU arm will receive the services based on mhGAP treatment protocols.
- TAU+Suicide Prevention Package (PSuPP) (Experimental): PCPs will receive all components of TAU. In addition, they receive an implementation package to optimize mhGAP siucide prevention delivery. The implementation package includes: [assessment optimization] systematic assessment training using systematized screening questions, an embedded decision-support tool, [risk management optimization] culturally adapted safety planning, and [follow up care optimization] a collaborative care protocol with Community Health Workers (CHWs) to support patient follow-up uptake and continued care. Participants in the PSuPP arm will receive all TAU services with aforementioned implementation strategies.
  Interventions: Behavioral: Suicide Prevention Package (PSuPP)

INTERVENTIONS:
Behavioral: Suicide Prevention Package (PSuPP) — Implementation package to optimize mhGAP siucide prevention delivery which includes: [assessment optimization] systematic assessment training using systematized screening questions, an embedded decision-support tool, [risk management optimization] culturally adapted safety planning, and [follow up care optimization] a collaborative care protocol with CHWs to support patient follow-up uptake and continued care.
  Arms: TAU+Suicide Prevention Package (PSuPP)

SUMMARY:
Suicide remains a major contributor to global mortality, with particularly high and persistent rates in low-resourced settings such as South Asia. In Nepal, ongoing integration of mental health services into primary care provides a critical opportunity to strengthen suicide risk assessment and management. Despite the scale-up of mhGAP training for primary care providers (PCPs), gaps remain in the systematic detection, referral, and follow-up of individuals at risk for suicide. There is an urgent need to enhance mhGAP implementation with strategies that address provider workload, stigma, and inequities within the health workforce.

Using experience-based co-design principles and RE-AIM this study will assess the feasibility and acceptability of integrating an implementation strategy package to optimize mhGAP suicide prevention delivery in Nepal's decentralized primary healthcare system. This clinical trial leverages deep collaboration with a community advisory board of individuals with lived experience of suicide throughout the trials' design, delivery and analysis.

This R34 will generate critical preliminary evidence on the feasibility, acceptability, and implementation of an integrated suicide prevention package within government primary care facilities in Nepal. The findings will inform the design and parameters of a future fully powered effectiveness trial, while aligning with Nepal's national suicide prevention strategy and advancing WHO and NIMH global mental health priorities.

ELIGIBILITY:
Inclusion Criteria:

Primary Care Providers

* Health workers with a prescribing license employed in government health facilities in Bagmati Province.
* Are between 21-65 years, per government health system criteria.
* Participants will be required to have competency in Nepali, be actively engaged in care provision within their health facility

Patients:

* Patient lives in the study site
* Is under the care of a PCP at a facility site.
* Patient meets any level of suicide risk based on mhGAP 2.0 criteria.
* Patients who have been treated for mental illness before or presently (expected in both groups).
* Speaks Nepali.
* Levels of Suicide Risk (as defined by mhGAP 2.0)

Exclusion Criteria:

Primary Care Providers

* Healthcare workers without proper government credentials will be excluded.
* Health workers who plan to migrate or who do not intend to stay in the study area for at least a year.

Patients:

* Patient requiring immediate hospitalization
* Unable to consent as determined by the diminished capacity tool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Percent intervention arm uptake to assess feasibility | 6 months
  Percent primary care providers (PCPs) that attend the implementation training. Feasibility will be defined as 70% or more uptake.
Percentage of interviews that hold themes | 6 months
  Qualitative feasibility acceptability data will be deemed acceptable if it demonstrates provider and patient perceptions of P-SuPP benefits to clinical care and mhGAP implementation and the absence of themes that suggest -SuPP is disruptive, unlikeable, and unacceptable. Acceptability will be assessed as the percentage of interviews that hold themes suggesting SuPP is disruptive, unlikeable, and unacceptable.
Percent retention to assess feasibility | 6 months
  Percent participants enrolled (PCPs and Patients) who complete the study of all enrolled. Feasibility is established as retention of at least 65% completion of 6 month follow up of patients and PCPs.
Structured checklist to assess fidelity | 6 months
  18-item structured checklist assessed in a standardized behavioral rehearsal to assess fidelity to the mhGAP suicide module protocol
Percent successful allocation procedures | 6 months
  Percent successful allocation procedures followed
Percent adherence to the randomization protocol | 6 months
  Percent adherence to the randomization protocol
Percent deviations to the randomization protocol | 6 months
  Percent deviations to the randomization protocol
Percent participants who completed all follow up measures | 6 months
  Percent participants who completed all follow up measures
Percent missing measure items per participant | 6 months
  Percent missing measure items per participant
Mean Beck Scale for Suicide Ideation (BSSI) score | Baseline; 3 months; 6 months
  Suicide ideation severity measured with BSSI. BSSI is a 19-item self-report instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviors, and plans to commit suicide during the past week. The first 19 items consist of three options graded are on a 3-point scale ranging from 0 to 2. These items are then summed to yield a total score, which ranges from 0 to 36. Higher scores indicate higher severity of suicide ideation. Assessed in patients only.

SECONDARY OUTCOMES:
Suicide Prevention Knowledge survey | Baseline, 3 months; 6 months
  The mhGAP knowledge survey includes 9 items related to suicide specific knowledge related to suicide risk presentation, management, and carer engagement aligned with the mhGAP suicide prevention protocol. Total score range XXXXX. Higher scores indicate more knowledge. Assessed in PCPs only.
Mean Self-Efficacy in Mental Health Care survey score | Baseline; 3 month; 6 month
  The mhGAP Self Efficacy is a self-administered measure assessing healthcare providers' confidence in assessing, diagnosing, and managing mental health conditions. Our adapted tool has 45 items across all domains and 8 items that focus specifically on suicide. Respondents select a range of responses between 1 and 5 with 1 feeling totally unable to do the domain and 5 feeling totally able to do the domain. Higher scores indicate higher self-efficacy. Assessed in PCPs only.
Mean Clinical Competency and Communication Skills (ENACT) score | Baseline; 6 months
  This is an observed role play with a trained rater to assess competence and interpersonal skills in delivering mental health interventions. The tool evaluates core competencies in psychological care delivery including: Communication, Emotional Engagement, Assessment, Social Relations, Planning and Process. communication skills, empathy, active listening, and patient engagement. Total score range 0-3. Higher scores indicate higher competence. Assessed in PCPs only.
Columbia Suicide Severity Rating Scale | Baseline; 3 months; 6 months
  The CSSRS asks about self-reported suicide attempt, aborted attempt, preparatory behavior, and interrupted attempt with "yes" or "no" questions branching format. Any positive responses to these behaviors will be coded as 'yes'. Behaviors are assessed at baseline as the past 3 months and lifetime and subsequent assessments have a window of the past three months. Participants will be categorized as low, medium or high risk based on their answers to specific questions. Assessed in patients only.
Mean Patient Health Questionnaire (PHQ-9) score | Baseline; 3 months; 6 months
  Depression measured with PHQ-9. PHQ-9 is a 9-item validated questionnaire. Each item asks about the frequency of specific depressive symptoms experienced over the past two weeks. The response options are scored from 0 to 3, indicating "not at all" to "nearly every day." The item scores are summed with total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Mean Suicide Cognitions Scale (SCS) score | Baseline; 3 months; 6 months
  The SCS includes 21 items that assess suicide-related cognitions, including negative expectations about the future, maladaptive self-perceptions, and emotional pain. The scale asks respondents to rate the extent to which they agree with experience specific suicide-related thoughts and beliefs. Responses are recorded on a Likert-type scale ranging from 1 to 5 from strongly disagree to strongly agree, and item scores are summed to produce a total score (21-105), with higher scores indicating greater severity of suicide-related cognitive distress. Assessed in patients only.
Suicide-Related Coping Scale (SRCS) - Internal Coping Skills | Baseline; 3 months; 6 months
  Assess suicide-related internal coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better internal coping). Assessed in patients only.
Suicide-Related Coping Scale (SRCS) - External Coping Skills | Baseline; 3 months; 6 months
  Assess suicide-related internal coping skills (7 items on 5-point scales; scores range from 0 to 28 with higher scores indicating better external coping). Assessed in patients only.
Mean Generalized Anxiety Disorder (GAD-7) score | Baseline; 3 months; 6 months
  Anxiety measured with GAD-7, a 7 item self report instrument that measures anxiety Items are scored on a 4-point scale, ranging from "not at all (0)" to "nearly everyday (3)". Item scores are summed with a total score ranging from 0 to 21: 0-4 Minimal anxiety; 5-9 Mild anxiety; 10-14 Moderate anxiety; 15-21 Severe anxiety. Assessed in patients only.
Mean Social Connectedness Scale score | Baseline; 3 months; 6 months
  The Social Connectedness Scale consists of 8 items that assess perceived sense of closeness, belonging, and connection with others. The scale consists of multiple items that ask respondents to rate their agreement on a scale of 1 to 5, with 1 indicating strong disagreement and 5 indicating strong agreement. Higher scores indicate higher social connection. Assessed in patients only.
Client Service Receipt Inventory to assess health service uptake | Baseline; 3 months; 6 months
  Percent services utilized will be assessed using the Client Services Receipt Inventory which measures use of health and social care services ranging from community delivered care from community health workers, to primary care services, to specialist services, and traditional health services. Assessed in patients only.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley K Hagaman, PhD, MPH, Principal Investigator — Yale School of Public Health
Locations (1):
- Primary care facilities, Dolakhā, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared through NIH designated data repositories consistent with data sharing under the NIH GDS policy. Clinical data of those research participants who will provide consent for sharing their data will be be included.